CLINICAL TRIAL: NCT04015102
Title: A Registry for Hereditary Cancer Risk Assessment and Genetic Testing Among Men With Prostate Cancer in the Community Urology Practice Setting
Brief Title: A Registry for Hereditary Cancer Risk Assessment and Genetic Testing
Status: Completed | Type: Observational
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Collaborators: Carolina Urologic Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: URO-012
Record Dates: First submitted 2019-06-26; First posted 2019-07-10 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer Patients; myRisk genetic testing
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood sample required for myRisk test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective registry will evaluate the feasibility and impact of implementing standard cancer family history review and guideline-aligned genetic testing for men diagnosed with Prostate Cancer in community urology practices nationwide.

DETAILED DESCRIPTION:
Genes linked to hereditary cancer syndromes have been associated with increased risk for prostate cancer (PrCa), earlier disease onset and increased disease aggressiveness.1,2 Ascertaining family cancer history and hereditary risk in men diagnosed with PrCa can help inform medical management decisions. Recently published National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology for Prostate Cancer (v3.2018)3 and Genetic/Familial High Risk Assessment: Breast and Ovarian (v2.2019)4 as well as the American Urological Association Guideline for Clinically Localized Prostate Cancer (2017)5 recommend appropriate counseling and genetic testing for men who are at increased hereditary cancer risk, based upon personal or family history. Genetic testing for patients with metastatic prostate cancer is now standard of care per NCCN Genetic/Familial High Risk Assessment: Breast and Ovarian (v2.2019) guidelines4. NCCN Prostate Cancer Guidelines (v3.2018)3 recommend obtaining a cancer-focused family history at diagnosis and consideration of germline genetic testing in multiple risk groups. Community urology practices can support guideline-aligned care by performing routine hereditary cancer risk assessment (HCRA), patient counseling and, when appropriate, genetic testing. This prospective registry will evaluate the feasibility and impact of implementing standard cancer family history review and guideline-aligned genetic testing for men diagnosed with PrCa in community urology practices nationwide.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years of age or older at time of enrollment
* Affected with Prostate Cancer (newly or previously diagnosed patients).
* Presents for a medical care visit and meets eligibility criteria for hereditary cancer genetic testing, based on personal and family cancer history and NCCN Practice Guidelines in Oncology (Prostate Cancer)
* Able to understand informed consent and agrees to participate in the registry.

Exclusion Criteria:

* Minors (younger than 18 years of age)
* Have had previous genetic testing for Hereditary Breast and Ovarian Cancer or Lynch Syndrome, or have previously undergone hereditary multi-gene, pan-cancer, or panel testing.
* Unable to provide routine clinical informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate Cancer patients, at least 18 years or older, who meet NCCN guidelines and eligibility criteria, who have a scheduled set appointment at Community Urology practices.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
To see how practical it would be to integrate a standard hereditary cancer risk assessment, patient counseling and genetic testing process into the community urology practice setting. | 18 weeks per site
  To see how practical it would be to integrate a standard hereditary cancer risk assessment , patient counseling and genetic testing process into the community urology practice setting. Also to evaluate the impact of the integrated process on provider and patient satisfaction. This registry will gather information to evaluate the feasibility of HCRA and genetic testing process integration in the Urology community practice setting. Analysis of the registry will compare historical pre-process integration data with post-integration data from the same providers within participating community Urology practices.

SECONDARY OUTCOMES:
To see what the proportion of community urology patients with PrCa is who complete each component of the HCRA, patient counseling and genetic testing process. | 18 weeks
  To see what the proportion of community urology patients with PrCa is who complete each component of the HCRA, patient counseling and genetic testing process. This registry will gather information to evaluate the feasibility of HCRA and genetic testing process integration in the Urology community practice setting. Analysis of the registry will compare historical pre-process integration data with post-integration data from the same providers within participating community Urology practices.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Shore, MD, Principal Investigator — Carolina Urologic Research Center
Locations (10):
- United States (10):
  - Arkansas Urology, Little Rock, Arkansas
  - Urology Associates of Central California, Fresno, California
  - Urologic Specialists of Northwest Indiana, Merrillville, Indiana
  - Comprehensive Urology, Royal Oak, Michigan
  - Comprehensive Urology, Waterford, Michigan
  - Associated Medical Professionals of New York, Syracuse, New York
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Oregon Urology Institute, Springfield, Oregon
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina